CLINICAL TRIAL: NCT05264415
Title: Interrupting the Intergenerational Transmission of Traumatic Stress: Identifying Parental Targets for Intervention by Looking Under the Skin
Brief Title: Intergenerational Transmission of Traumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nastassia Hajal, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KHD097277A; 1K08HD097277-01A1 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2022-03-03 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Stress, Psychological; Stress Disorders, Traumatic; Emotion Regulation; Behavior, Child; Emotional Stress; Trauma, Psychological; Anxiety; Depression; Coping Skills; Parent-Child Relations; Parenting
Keywords: Resilience; Families; Parents; Children; Preschooler; Intervention
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Traumatic; Emotional Regulation; Child Behavior; Psychological Trauma; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families Over-Coming Under Stress-Early Childhood Program (FOCUS-EC) (Experimental): FOCUS-EC is a trauma-informed, family-level, skill building program that provides developmental guidance, parent education, and key resilience skills that promote positive individual and family coping (including emotional regulation, problem solving, goal setting, communication, and management of trauma & loss reminders), which foster parent-child and family cohesion. It is delivered in approximately 8 weekly sessions (including approximately six 60-minute sessions with parent/caregivers only, and two 30-60 minute sessions with children and parent/caregivers together). Each session is structured with a check-in, review of the previous week's "home activity," new skills-based activity and discussion, selection of a new "home activity," and a closing check-out. FOCUS-EC promotes parenting skills and more cohesive family relationships in two key phases: 1) creating a family timeline and 2) enhancing parent-child interactions.
  Interventions: Behavioral: Families OverComing Under Stress (FOCUS) for Early Childhood (FOCUS-EC)
- Parenting Education Website (Active Comparator): The Parenting Education Website includes information and high-quality parenting resources covering topics such as typical child development, common child reactions to family stress and transitions, play, positive parenting strategies, and the importance of self-care.
  Interventions: Other: Parenting Education Website

INTERVENTIONS:
Behavioral: Families OverComing Under Stress (FOCUS) for Early Childhood (FOCUS-EC) — Trauma-informed, family-centered, skill-building preventive intervention for families with preschool-aged children.
  Arms: Families Over-Coming Under Stress-Early Childhood Program (FOCUS-EC)
Other: Parenting Education Website — A website providing parenting education resources in four primary domains relevant for families with preschool-aged children (parenting, child development, transitions, and self-care).
  Arms: Parenting Education Website

SUMMARY:
Millions of U.S. parents have experienced trauma, putting them at risk for maladaptive parenting practices, which then confer vulnerabilities to their children. This study aims to enhance understanding of how parental emotional dysregulation associated with traumatic stress impedes effective parenting. The study employs neurophysiological methods (electroencephalogram; EEG) to address some of the challenges inherent in the study of emotion (particularly in trauma-exposed individuals) and to identify potential biomarkers of traumatic stress and response to intervention.

DETAILED DESCRIPTION:
This research study consists of a randomized controlled trial of 60 families of preschool-aged children in which a parent/caregiver has their own history of childhood interpersonal trauma or loss.

Parent/caregiver participants and their preschool-aged child will participate in two phases of assessment (baseline/Time 1 and follow-up/Time 2). Each phase of assessment will include parent/caregiver participant completion of self-report questionnaire measures, a parent-child interaction task (which will be video-recorded for later behavioral coding) and a parent EEG assessment. After the Time 1 (T1) assessments, participants will be randomized to either the FOCUS-Early Childhood Program group (n = 30; experimental group) or the parent education curriculum website group (n = 30; active comparator group).

The T2 assessment phase will begin at 3-months post-baseline. The FOCUS-EC Program is an 8-week program, so families should have completed the program by 3 months post-baseline. In the event that a family that was randomized to the FOCUS-EC Program group has not completed the program by the 3-month mark, the T2 assessment will be initiated once the program has been completed (up to 6 months post-baseline).

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver (must be legal guardian) of a 3- to 6-year-old child
* Child must cohabitate with the parent/caregiver
* Parent/caregiver participant must have experienced some form of interpersonal trauma during their own childhood (e.g., abuse, neglect, witnessing domestic violence)
* Parent/caregiver must be English-speaking
* Parent/caregiver must have access to internet and Webcam

Exclusion Criteria:

* Does not meet inclusion criteria
* Parent/legal guardian does not want the child to participate in the study
* Significant neurological disorder (included in pre-screening protocol)
* Active psychosis/mania (as assessed by staff)
* Significant child developmental delays (as assessed by staff)

Families excluded from the study will be provided with a list of online and/or community resources.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Change in observed parenting behaviors during standardized parent-child interaction tasks | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  Coded based on previously established parent-child behavioral coding systems (Deater-Deckard, 2000; Deater-Deckard, Pylas, & Petrill, 1997; Dix et al., 2004; Murphy, Boyd-Soissan, et al., 2017), including codes for positive parenting behaviors (e.g., praise, sensitivity, positive affect expressions), negative parenting behaviors (e.g., criticism, intrusiveness, harshness, negative affect expressions), and responses to children's negative emotion expressions (e.g., emotion coaching, validation, suppression, minimization).
Change in self-reported parenting behaviors as measured by the Multidimensional Assessment of Parenting Scale (MAPS) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Multidimensional Assessment of Parenting Scale (MAPS) is a self-report questionnaire of parenting behaviors. This study will administer the 30 items corresponding to subscales that represent the following aspects of parenting behavior:
  * proactive parenting
  * positive reinforcement
  * warmth
  * supportiveness
  * hostility
  * lax control
  The scale is scored such that higher scores indicate a higher degree of that type of parenting (e.g., higher scores on the positive reinforcement subscale indicate greater use of positive reinforcement).
  Each subscale:
  Minimum possible score: 1 Maximum possible score: 5
Change in posttraumatic stress disorder symptoms as measured by the Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5) is a well-established, 20-item questionnaire of posttraumatic stress symptoms. Higher scores indicate higher levels of posttraumatic stress symptoms.
  Minimum possible score: 0 Maximum possible score: 80

SECONDARY OUTCOMES:
Change in Emotion Regulation Questionnaire (ERQ) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report questionnaire that assesses emotion regulation strategies of cognitive reappraisal and expressive suppression, with higher scores indicating greater use of those strategies.
  Minimum possible score: 1 Maximum possible score: 7
Change in Parental Feelings Inventory (PFI) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Parental Feelings Inventory (PFI) is a 31-item self-report questionnaire that assesses parents' experience of specific emotions in the parenting context (Bradley et al., 2013). Higher scores represent greater experience of each type of emotion in the parenting role within the past month.
  Minimum possible score: 1 Maximum possible score: 7
Change in Parental Emotion Regulation Inventory-2 (PERI-2) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Parental Emotion Regulation Inventory-2 (PERI-2) is a self-report questionnaire that assesses coping and emotion regulation strategies used within the parenting context (Lorber et al., 2017). The scale includes 23 items corresponding to subscales that represent the following aspects of emotion regulation:
  * reappraisal
  * suppression
  * capitulation
  * escape
  The scale is scored such that higher scores indicate a higher degree of that type of strategy (e.g., higher scores on the reappraisal subscale indicate greater use of reappraisal).
  Minimum possible score: 1 Maximum possible score: 7
Change in Coping with Children's Negative Emotions Scale (CCNES) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Coping with Children's Negative Emotions Scale (CCNES) is an 82-item self-report questionnaire that assesses parents' responses to children's displays of negative emotions (e.g., expressive encouragement, problem solving, punishment, minimization). Higher scores reflect higher use of that type of response (e.g., higher score on expressive encouragement subscale indicates higher use of expressive encouragement responses).
  Minimum possible score: 1 Maximum possible score: 7
Change in Patient Health Questionnaire-8 (PHQ-8) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Patient Health Questionnaire-8 (PHQ-8) is a well-established, 8-item scale of depression symptoms, with higher total scores indicating higher levels of depression symptoms.
  Minimum possible score: 0 Maximum possible score: 24
Change in Generalized Anxiety Disorder-7 Questionnaire (GAD-7) | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Generalized Anxiety Disorder-7 Questionnaire (GAD-7) is a well-established, 7-item scale of anxiety symptoms, with higher total scores indicating higher levels of anxiety symptoms.
  Minimum possible score: 0 Maximum possible score: 21
Change in Parenting Stress Index-Short Form 4 | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Parenting Stress Index-Short Form 4 (PSI-SF) is a 36-item self-report questionnaire of three dimensions of parenting stress (parental distress, parent-child dysfunctional interaction, and difficult child). Higher scores indicate higher levels of parenting stress.
  Subscales:
  Minimum possible score: 12 Maximum possible score: 60
  Total Score:
  Minimum possible score: 36 Maximum possible score: 180
Change in Eyberg Child Behavior Inventory | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Eyberg Child Behavior Inventory (ECBI) is a 36-item parent/caregiver-report questionnaire measure of children's behavior problems that obtains information about the frequency of problem behaviors (Intensity subscale; higher scores indicate greater intensity) and whether or not the behavior is problematic for the parent (Problem subscale; higher scores indicate greater problem).
  Behavior intensity:
  Minimum possible score: 36 Maximum possible score: 252
  Problem behavior:
  Minimum possible score: 0 Maximum possible score: 36
Change in Preschool Feelings Checklist | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Preschool Feelings Checklist is a 16-item parent/caregiver-report questionnaire measure of children's depressive symptoms. Higher scores indicate higher depression symptoms.
  Minimum possible score: 0 Maximum possible score: 16
Change in Spence Child Anxiety Scale - Preschool Version | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Spence Child Anxiety Scale - Preschool Version is a 34-item parent/caregiver-report questionnaire measure of children's anxiety symptoms. Higher scores indicate higher anxiety symptoms.
  Minimum possible score: 0 Maximum possible score: 112

OTHER OUTCOMES:
Change in electroencephalography (EEG)-measured cortical alpha asymmetry | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  EEG will be used to examine parent/caregiver alpha asymmetry in the frontal and parietal cortices during several tasks:
  - Resting baseline tasks:
  1. 4 minutes of eyes open
  2. 4 minutes of eyes closed
     - Explicit emotion tasks:
  3. Participants passively view images of children
  4. Participants are asked to pay attention to and modulate their emotions while viewing images of children
  5. Participants engage in a task of executive functioning (Go/No-Go paradigm) that uses photos of children's facial emotion expression as stimuli
     - Implicit emotion task:
  6. Participants view photos of children's facial emotion expressions and are asked to categorize them by gender
Change in electroencephalography (EEG)-measured cortical functional connectivity | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  EEG will be used to examine parent/caregiver functional connectivity between the frontal and parietal cortices during several tasks:
  - Resting baseline tasks:
  1. 4 minutes of eyes open
  2. 4 minutes of eyes closed
     - Explicit emotion tasks:
  3. Participants passively view images of children
  4. Participants are asked to pay attention to and modulate their emotions while viewing images of children
  5. Participants engage in a task of executive functioning (Go/No-Go paradigm) that uses photos of children's facial emotion expression as stimuli
     - Implicit emotion task:
  6. Participants view photos of children's facial emotion expressions and are asked to categorize them by gender
Change in Parent Reflective Functioning Questionnaire | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Parent Reflective Functioning Questionnaire is a self-report questionnaire measure of parental reflective functioning. The questionnaire consists of 18 items corresponding to subscales that represent the following aspects of reflective functioning:
  * Pre-mentalizing
  * Certainty about Mental States
  * Interest and Curiosity in Mental States
  The scale is scored such that higher scores indicate a higher degree of that type of reflective functioning (e.g., higher scores on the Certainty about Mental States subscale indicate greater certainty about infant mental states).
  Minimum possible score: 1 Maximum possible score: 7
Change in Perth Alexithymia Questionnaire | Time 1 (baseline assessment) and Time 2 (3-months post-baseline)
  The Perth Alexithymia Questionnaire is a 24-item self-report questionnaire measure of alexithymia, with higher scores indicating higher levels of alexithymia.
  Minimum possible score: 24 Maximum possible score: 168

CONTACTS AND LOCATIONS:
Overall Officials: Nastassia Hajal, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States